CLINICAL TRIAL: NCT05073536
Title: Feasibility of Mini-sized Magnetically Controlled Capsule Endoscopy in Visualization of UGI and Small Bowel: a Randomized Controlled Clinical Trial
Brief Title: Mini-sized MCE for Better Examination of UGI and Small Bowel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: mini-MCE
Record Dates: First submitted 2021-09-17; First posted 2021-10-11 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Capsule Endoscopy
Keywords: magnetically controlled capsule endoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mini-sized MCE (Experimental): Participants in this group underwent examination of mini-sized MCE.
  Interventions: Device: mini-sized MCE
- normal-sized MCE (Other): Participants in this group underwent examination of normal-sized MCE.
  Interventions: Device: normal-sized MCE

INTERVENTIONS:
Device: mini-sized MCE — Enrolled participants were randomly allocated into the normal-sized MCE group or mini-sized MCE group in a 1:1 ratio.
  Arms: mini-sized MCE
Device: normal-sized MCE — Enrolled participants were randomly allocated into the normal-sized MCE group or mini-sized MCE group in a 1:1 ratio.
  Arms: normal-sized MCE

SUMMARY:
A mini-sized MCE highlighted with a diameter of 9.5mm, a length of 24.5mm, and a weight of 3.0g has been developed. This new type of MCE is approximately 0.6 times the conventional MCE (27mm*11.8mm) in volume and weight, and it is the smallest CE among all the reported capsules. Thus, this pilot study was conducted to clarify whether the mini-sized MCE can further optimize the process of swallowing the capsule and to verify whether the smaller size of the capsule will have influence on the examination procedure of the upper gastrointestinal tract and small intestine.

DETAILED DESCRIPTION:
Magnetically controlled capsule endoscopy (MCE), with equally favorable diagnostic accuracy as conventional endoscopy, has become a painless noninvasive diagnostic modality in clinical practice. The more than 8 hours battery life of the MCE enables a further examination of the small bowel. In addition, it has been demonstrated that magnetic steering of capsule endoscopy improves the completion rate of small bowel examination by facilitating passage of the capsule through the pylorus, which further supported MCE as a practical modality for examination of both the stomach and small bowel. Previous studies have confirmed the great safety and efficacy of MCE for examination of patients with high-risk factors for standard gastroscopy, those long-time taking aspirin, aging patients and children.

However, this technique still has some limitations in clinical practice. Due to the large size of the capsule, some patients may be difficult to swallow the capsule, especially in children. A clinical trial reported that a certain number of children with ages ranging from 6 to 14 years fail to swallow the MCE by themselves for its big size (27mm*11.8mm). During the examination procedure of small bowel capsule endoscopy, measuring 26*11mm, in those under 10 years old of age, up to 87% of patients are unable to swallow the capsule. In adolescents, it is reported that more than one-third of patients have difficulties with swallowing standard size tablets. In addition, serious complications, such as aspiration of the capsule, often occur in the elderly who need more efforts to swallow the capsule. For those at any age unable or unwilling to swallow a capsule, endoscopic placement is required to deliver the capsule to the stomach or directly the duodenum. However, this procedure greatly increases patient's discomfort, examination costs and increase the risk associated with the endoscopic procedure, anesthesia. Thus, it is of great importance to make the capsule endoscopy easier to swallow in both children and adolescents.

Therefore, a mini-sized MCE highlighted with a diameter of 9.5mm, a length of 24.5mm, and a weight of 3.0g has been developed. This new type of MCE is approximately 0.6 times the conventional MCE (27mm*11.8mm) in volume and weight, and it is the smallest CE among all the reported capsules. Thus, this pilot study was conducted to clarify whether the mini-sized MCE can further optimize the process of swallowing the capsule and to verify whether the smaller size of the capsule will have influence on the examination procedure of the upper gastrointestinal tract and small intestine.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18.
* Scheduled to undergo a capsule endoscopy for both stomach and small bowel.
* Signed the informed consents before joining this study.

Exclusion Criteria:

* Dysphagia or symptoms of gastric outlet obstruction
* Known or suspected GI obstruction, stenosis, or fistula
* History of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy
* Implanted pacemaker, except the pacemaker is compatible with MRI
* Other implanted electromedical devices or magnetic metal foreign bodies
* Pregnancy or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
the difficulty score for swallowing the capsule | 6 months
  The primary outcome was the difficulty score for swallowing the capsule, which was assessed on a visual analog scale ranging from 0 (very easy with no nausea) to 10 (very difficult or with severe nausea)
the time required to swallow the capsule | 6 months
  The capsule swallowing time was defined as the time between the first mouth image and the first esophageal image.
the success rate for swallowing the capsule at the first attempt | 6 months
  If the patient swallowed the capsule directly with a sip of water at the first attempt, it was defined as a success for swallowing the capsule at the first attempt; if the capsule entered the esophagus after several swallowing attempts or with endoscopic placement, it was defined as a failure.

SECONDARY OUTCOMES:
the number of images captured for Z-line and quadrants of the Z-line | 6 months
  Visualization of the esophagus indicated by the number of images captured for Z-line and how many quadrants of the Z-line were observed.
Visualization score of the gastric mucosa | 6 months
  To objectively evaluate the complete visualization of the gastric mucosa in the 6 anatomic landmarks (cardia, fundus, body, angulus, antrum, and pylorus), a 3-point grading scale was used: 1, poor (<70% of the mucosa was observed), 2, fair (70%-90% of the mucosa was observed), and 3, good (>90% of the mucosa was observed).
Visualization of the small bowel | 6 months
  Visualization of the small bowel was determined by the small bowel complete examination rate.
Difficulty score of swallowing the capsule | 1 month
  To evaluate the difficulty score of swallowing the capsule. After the examination, the patient was asked to complete a questionnaire. A visual analogue scale ranging from 0 (easy with no nausea) to 10 (very difficult or with sever nausea) was used to evaluate the degree of difficulty of swallowing the capsule.
Gastrointestinal transit time | 1 month
  Examination-related parameters included esophageal transit time (ETT), gastric examination time (GET), gastric transit time (GTT), pylorus transit time (PTT), small bowel transit time (SBTT). ETT is defined as the time between the first esophageal image and the first gastric image. GTT is defined as the time between the first gastric image and the first duodenal image. GET is defined as the time for examination of gastric primary anatomic landmarks twice. PTT is defined as the time between the first pyloric image and the first duodenal image. SBTT is defined as the time between the first duodenal image and the first cecal image.
Detection rate of lesions | 1 month
  The detection rate of lesions in different digestive part (esophagus, stomach, duodenum, small intestine) found by mini-sized MCE and normal-sized MCE.
Safety of mini-sized MCE procedure:presence of any adverse events during mini-sized MCE procedure will be recorded | 1 month
  presence of any adverse events during mini-sized MCE procedure will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Professor, Principal Investigator — Changhai Hospital,Shanghai,China
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Liao Z, Zou W, Li ZS. Clinical application of magnetically controlled capsule gastroscopy in gastric disease diagnosis: recent advances. Sci China Life Sci. 2018 Nov;61(11):1304-1309. doi: 10.1007/s11427-018-9353-5. Epub 2018 Oct 18. PMID 30367341
- [Background] Jiang X, Pan J, Li ZS, Liao Z. Standardized examination procedure of magnetically controlled capsule endoscopy. VideoGIE. 2019 May 30;4(6):239-243. doi: 10.1016/j.vgie.2019.03.003. eCollection 2019 Jun. No abstract available. PMID 31194028
- [Background] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825
- [Background] Hu J, Wang S, Ma W, Pan D, Sun S. Magnetically controlled capsule endoscopy as the first-line examination for high-risk patients for the standard gastroscopy: a preliminary study. Scand J Gastroenterol. 2019 Jul;54(7):934-937. doi: 10.1080/00365521.2019.1638446. Epub 2019 Jul 22. PMID 31328998
- [Background] Nuutinen H, Kolho KL, Salminen P, Rintala R, Koskenpato J, Koivusalo A, Sipponen T, Farkkila M. Capsule endoscopy in pediatric patients: technique and results in our first 100 consecutive children. Scand J Gastroenterol. 2011 Sep;46(9):1138-43. doi: 10.3109/00365521.2011.584900. Epub 2011 May 26. PMID 21615227
- [Background] Patel A, Jacobsen L, Jhaveri R, Bradford KK. Effectiveness of pediatric pill swallowing interventions: a systematic review. Pediatrics. 2015 May;135(5):883-9. doi: 10.1542/peds.2014-2114. PMID 25896843
- [Background] Dan T, Dandan S, Enqiang L. Aspiration of a Magnetically Controlled Capsule Endoscopy. Gastroenterology. 2023 May;164(6):e30-e31. doi: 10.1053/j.gastro.2019.04.006. Epub 2019 Apr 11. No abstract available. PMID 30981792
- [Derived] Jiang X, Qiu XO, Li Z, Pan J, Peng C, Zuo XL, Liao Z, Li ZS. Small-sized versus standard magnetic capsule endoscopy in adults: a two-center, double-blinded randomized controlled trial. Endoscopy. 2023 Jan;55(1):52-57. doi: 10.1055/a-1881-4369. Epub 2022 Jul 12. PMID 35820437